CLINICAL TRIAL: NCT05325970
Title: Clinical Registry of Long-Term Dental Outcomes in Head and Neck Cancer Patients (ORARAD II)
Brief Title: Clinical Registry of Long-Term Dental Outcomes in Head and Neck Cancer Patients
Acronym: ORARAD II
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); University of Minnesota (Other); UConn Health (Other); University of Pennsylvania (Other); Brigham and Women's Hospital (Other); NYU Langone Health (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00091445; U01DE022939 (NIH); Pro00060322 (Other: Atrium Health)
Record Dates: First submitted 2022-03-25; First posted 2022-04-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Head and Neck Cancer; Dental Diseases; Osteoradionecrosis
Keywords: dental outcomes; cancer; registry
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatognathic Diseases; Osteoradionecrosis; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohorts Interventions Patients receiving head and neck RT

SUMMARY:
The current study (ORARAD II) will examine participants of the original cohort for a visit roughly 7 years after the start of RT. The primary outcomes will be the 7-year rate of dental caries, periodontal disease, tooth loss, osteoradionecrosis and salivary flow.

DETAILED DESCRIPTION:
This is a prospective cohort study to document long-term dental and other oral outcomes in patients who receive external beam and modern radiation therapy (RT) modalities with curative intent, as part of clinical care for a head and neck cancer. Five hundred and seventy-two participants were enrolled in the original study, ORARAD, which included a baseline oral examination prior to the start of radiation therapy and follow-up examinations and data collection at six-month intervals up to 2 years after the start of RT. The current study (ORARAD II) will examine participants of the original cohort for a visit roughly 7 years after the start of RT. The primary outcomes will be the 7-year rate of dental caries, periodontal disease, tooth loss, osteoradionecrosis and salivary flow.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the original ORARAD study
* Willing to participate and comply with all study procedures

Exclusion Criteria:

* Anything that would place the participant at increased risk or preclude the participant's full compliance with or completion of the study (e.g., unable to obtain consent or unable to tolerate an oral examination).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be offered to all living ORARAD participants approximately 7 years post-RT. Persons of all races and ethnicities and both females and males will thus be eligible for this study. Because participants will be drawn solely from the participants in the original ORARAD, the racial/ethnic composition of the study population at each center will be determined by the composition of those enrolled in the original ORARAD, which has been documented elsewhere. Since there is no evidence to suggest that dental outcomes in head and neck cancer patients are affected by gender, this expected unequal gender distribution of study participants will not affect the scientific validity of the study. Individuals who meet the eligibility criteria will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Dental Caries | 7 years
  Dental caries will be ascertained through the examination parameters outlined by NHANES, and the results of this examination with be used to calculate DMFS scores.
Bleeding on probing is documented (yes/no) (Periodontal Measure 1) | 7 years
  Bleeding on probing is documented (yes/no) and a percentage of "yes" responses will be calculated.
Clinical attachment loss (CAL) (Periodontal Measure 2) | 7 years
  Clinical attachment loss (CAL) measured in mm
Pocket depth (Periodontal Measure 3) | 7 years
  Pocket depth measured in mm
Tooth Loss | 7 years
  "Tooth loss" will be defined as a dental extraction that has been performed or recommended. Change in number of teeth throughout the duration of the study will be documented.
Exposed intraoral bone | 7 years
  Exposed intraoral bone is documented clinically by a trained clinical examiner and assessed based on a visual examination of the area, documenting the related tooth numbers or area and the following clinical signs: pain, swelling, induration, sequestrum, thin skin and/or beard loss (i.e. tissue hypoxia), evidence of pathologic fracture, tooth mobility, altered sensation in the affected area. The percentage of patients experiencing exposed bone, their recovery rates, and percent experiencing the signs will be calculated.
Salivary flow | 7 years
  Salivary flow is measured by the whole stimulated salivary flow rate. Changes in the rate and any association with other outcomes (e.g., caries) will be calculated.

SECONDARY OUTCOMES:
Trismus measurements in mm | 7 years
  Change in mouth opening are documented in mm
7-year use of fluoride | 7 years
  Patients complete a questionnaire on use of fluoride (other than over the counter toothpaste), type, and frequency. Percent compliance with fluoride use and change in fluoride use will be calculated.
Compliance with brushing/flossing | 7 years
  Patients complete a questionnaire on frequency of brushing and flossing. Percent compliance with brushing and flossing guidelines (2x per day according to evidence-based professional guidelines) and change in compliance will be calculated.
Changes in RT-specific quality of life measures | 7 years
  Patients complete a likert scale questionnaire on 10 quality of life measures based on the European Organization for Research and Treatment of Cancer questionnaire. Ten individual question items were scored on a four-point scale indicating level of difficulty with daily tasks (1=not at all; 2=a little; 3=quite a bit; 4=very much).
Change in pain scores | 7 years
  Patients complete a likert scale questionnaire on pain levels during 8 daily activities rating their pain from no pain (0) to the worst pain imaginable (5) based on the European Organization for Research and Treatment of Cancer questionnaire.
Mortality | 7 years
Cancer recurrence | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael T. Brennan, DDS, MHS, Principal Investigator — Wake Forest University Health Sciences; Rajesh V. Lalla, DDS, PhD, Principal Investigator — UConn Health
Locations (6):
- United States (6):
  - University of Connecticut Health Center - School of Dental Medicine, Farmington, Connecticut
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - New York University - College of Dentistry, New York, New York
  - University of North Carolina School of Dentistry, Chapel Hill, North Carolina
  - University of Pennsylvania School of Dental Medicine, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
PI will share deidentified data , no other documents, upon reasonable request
Supporting Information: Study Protocol
Time Frame: immediately after publication, no expiration
Access Criteria: send request to either Dr. Brennan (mike.brennan@atriumhealth.org) or Dr. Rajesh Lalla (lalla@uconn.edu).